CLINICAL TRIAL: NCT03236194
Title: Ancillary Microbiome Collection From Mother/Infant Pairs During First Year of Life
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Collaborators: Penn State University (Other)
Responsible Party: Principal Investigator, Ian M. Paul, MD, Professor of Pediatrics and Public Health Sciences Chief, Division of Academic General Pediatrics Vice Chair of Clinical Affairs, Department of Pediatrics, Milton S. Hershey Medical Center
Other Study IDs: PRAMS034493EP
Record Dates: First submitted 2017-07-25; First posted 2017-08-01 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Infant Development

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — microbiome samples from mother and infant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators will be studying the development of the microbiome over the first year after birth in light of various environmental influences - e.g. mode of delivery, diet (and diet changes), antibiotic exposure, GERD medication exposure.

DETAILED DESCRIPTION:
Microbiome samples will be collected from mother/infant pairs during post-natal hospital stay through the first year of life. Investigators will perform statistical analyses to test the hypotheses (1) that there is an association between the developing oral and gut microbiomes, and (2) that they interact in affecting childhood obesity.

This study relates to the INSIGHT study (NCT01167270) and its last outcome measure; exploring oral and gut microbiome collected from that study's second born participants.

ELIGIBILITY:
Inclusion Criteria:

1. full-term infant (> 36 0/7 weeks gestational age) without significant morbidity
2. nursery/NICU/maternity stay of 7 days or less
3. participant children can be (but do not have to be) twins
4. English speaking mother
5. care provided at an HMC affiliated clinic
6. a working telephone number

Exclusion Criteria:

1. prenatal ultrasound presence of intrauterine growth retardation (IUGR)
2. infant birth weight <2250 grams
3. presence of a congenital anomaly or neonatal condition that significantly affects a newborn's feeding (e.g. cleft lip, cleft palate, metabolic disease)
4. any major maternal morbidities and/or pre-existing condition that would affect postpartum care or her ability to care for her newborn such as cancer, multiple sclerosis, lupus, etc.
5. plan for newborn to be adopted
6. plan to move from Central Pennsylvania within 1 year
7. have 2 older siblings in INSIGHT/SIBSIGHT (NIH funded study related to this ancillary study)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy full-term mothers and infants delivering at the Penn State Milton S Hershey Medical center.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Microbiome outcome | birth to 1 year
  Microbiome diversity within individuals (how gut and oral microbiomes are similar or different) and between individuals

SECONDARY OUTCOMES:
Genetic variation | birth to 1 year
  Associations between genetic variation and microbiome diversity
Genetic variation | birth to 1 year
  Genetic variation as it relates to growth outcomes

CONTACTS AND LOCATIONS:
Locations (1):
- Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Gomez A, Nelson KE. The Oral Microbiome of Children: Development, Disease, and Implications Beyond Oral Health. Microb Ecol. 2017 Feb;73(2):492-503. doi: 10.1007/s00248-016-0854-1. Epub 2016 Sep 14. PMID 27628595
- [Background] Gritz EC, Bhandari V. The human neonatal gut microbiome: a brief review. Front Pediatr. 2015 Mar 5;3:17. doi: 10.3389/fped.2015.00017. eCollection 2015. PMID 25798435
- [Background] Chu DM, Ma J, Prince AL, Antony KM, Seferovic MD, Aagaard KM. Maturation of the infant microbiome community structure and function across multiple body sites and in relation to mode of delivery. Nat Med. 2017 Mar;23(3):314-326. doi: 10.1038/nm.4272. Epub 2017 Jan 23. PMID 28112736
- [Background] Backhed F, Roswall J, Peng Y, Feng Q, Jia H, Kovatcheva-Datchary P, Li Y, Xia Y, Xie H, Zhong H, Khan MT, Zhang J, Li J, Xiao L, Al-Aama J, Zhang D, Lee YS, Kotowska D, Colding C, Tremaroli V, Yin Y, Bergman S, Xu X, Madsen L, Kristiansen K, Dahlgren J, Wang J. Dynamics and Stabilization of the Human Gut Microbiome during the First Year of Life. Cell Host Microbe. 2015 Jun 10;17(6):852. doi: 10.1016/j.chom.2015.05.012. Epub 2015 Jun 10. No abstract available. PMID 26308884